CLINICAL TRIAL: NCT01073306
Title: A Phase I Evaluation of the Safety and Immunogenicity of rDEN2/4 Δ30(ME) Dengue Serotype 2 Vaccine Given at 10^1 PFU in Healthy Flavivirus-naïve Adult Subjects
Brief Title: Safety and Immune Response to an Investigational Dengue Type 2 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 254; #20081980 (Other: WIRB Protocol Number)
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Dengue Virus
Keywords: Vaccine; Dengue Hemorrhagic Fever
MeSH Terms: conditions — Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dengue Virus Subtype 2 Vaccine (Experimental): Participants will receive a single dose of investigational vaccine for dengue virus subtype 2.
  Interventions: Biological: Investigational Vaccine for Dengue Virus Subtype 2
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo vaccine.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Investigational Vaccine for Dengue Virus Subtype 2 — Subcutaneous injection in upper arm of vaccine at dose of 10 plaque-forming units (PFU)
  Other Names: rDEN2/4Δ30
  Arms: Dengue Virus Subtype 2 Vaccine
Other: Placebo — Subcutaneous injection of placebo
  Arms: Placebo

SUMMARY:
Dengue viruses can cause dengue fever and other serious health conditions, primarily affecting people living in tropical regions of the world. This study will test whether a vaccine developed to prevent infection with dengue virus type 2 causes a response in people's immune system and is safe.

DETAILED DESCRIPTION:
Dengue viruses cause approximately 50 million cases of dengue fever and 1.5 million cases of the more severe diseases dengue hemorrhagic fever (DHS) and dengue shock syndrome (DSS) every year. There are four subtypes of the virus, and infection with one offers no protection from infection by the others. In fact, most cases of DHS and DSS occur in people infected by more than one subtype. In areas of the world where multiple subtypes of dengue are common, vaccines must be developed against each of the subtypes of dengue virus. This study will examine the safety and immune response of an investigational vaccine for preventing dengue virus type 2.

Participation in this study will last about 6 weeks. Participants will be randomly assigned to be injected with either the investigational study vaccine or a placebo. Participants will have a five in six chance of receiving the vaccine. The first study visit will take place on the vaccination day, on which participants will undergo a physical examination, blood draw, and pregnancy test and then receive the vaccine. Participants will be given a thermometer and temperature card and be told to record their temperatures three times per day for 16 days after vaccination. Participants will come to follow-up visits every other day for the 16 days after vaccination and then 3, 4, and 6 weeks after vaccination (Days 21, 28, and 42). Assessments completed during these visits will include a questionnaire about how the participant is feeling, pregnancy test, review of temperature cards, blood draw, and physical exam. Blood drawn will be analyzed to check participants' health, determine the amount of vaccine and antibodies in the blood, test markers in white blood cells and genes, and look for proteins that are important for fighting dengue infection.

ELIGIBILITY:
Inclusion Criteria:

* Good general health as determined by physical examination, laboratory screening, and review of medical history
* Available for the duration of the study, approximately 6 weeks post-vaccination
* Female participants of childbearing potential must be willing to use effective contraception for the duration of the trial

Exclusion Criteria:

* Currently breastfeeding or pregnant
* Exhibits evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Presence of a behavioral, cognitive, or psychiatric disease that affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Has screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in protocol
* Presence of any condition that would jeopardize the safety or rights of the participant or would render the participant unable to comply with the protocol
* Significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Presence of severe asthma, defined as requiring emergency room visit or hospitalization within the last 6 months
* Presence of HIV infection, determined by screening and confirmatory assays
* Presence of hepatitis C virus (HCV) infection, determined by screening and confirmatory assays
* Presence of hepatitis B virus (HBV) infection, determined by hepatitis B surface antigen (HBsAg) screening
* Presence of any known immunodeficiency syndrome
* Uses anticoagulant medications
* Has used corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination. An immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone or equivalent per day for greater than or equal to 14 days.
* Has received a live vaccine within 28 days or a killed vaccine within 14 days prior to vaccination or anticipates receipt of any vaccine during the 42 days following vaccination
* Has no spleen
* Has received blood products within the past 6 months, including transfusions or immunoglobulin, or anticipates receipt of any blood products or immunoglobulin during the 42 days following vaccination
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis, West Nile virus)
* Has received a flavivirus vaccine (licensed or experimental)
* Anticipates receipt of any investigational agent in the 42 days before or after vaccination
* Has definite plans to travel to a dengue endemic area during the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of vaccine, as assessed by neutralizing antibody titers | Measured at 4 and 6 weeks after vaccination
Safety of vaccine, as assessed by the frequency of vaccine-related adverse events (AEs), graded by severity | Measured throughout study
Number of vaccinees infected with this dengue virus subtype 2 (DEN2) candidate vaccine, as defined by either recovery of vaccine virus from the blood of vaccinated participants and/or by seroconversion to DEN2 | Measured at Days 28 and 42

SECONDARY OUTCOMES:
Frequency, quantity, and duration of viremia | Measured after vaccination
Comparison of infectivity rates, safety, and immunogenicity of a single dose of DEN2 vaccine from this trial to those variables on previous trials | Measured at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Project SAVE, Center for Immunization Research, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Blaney JE Jr, Durbin AP, Murphy BR, Whitehead SS. Development of a live attenuated dengue virus vaccine using reverse genetics. Viral Immunol. 2006 Spring;19(1):10-32. doi: 10.1089/vim.2006.19.10. PMID 16553547
- [Background] Durbin AP, McArthur JH, Marron JA, Blaney JE, Thumar B, Wanionek K, Murphy BR, Whitehead SS. rDEN2/4Delta30(ME), a live attenuated chimeric dengue serotype 2 vaccine is safe and highly immunogenic in healthy dengue-naive adults. Hum Vaccin. 2006 Nov-Dec;2(6):255-60. doi: 10.4161/hv.2.6.3494. Epub 2006 Nov 5. PMID 17106267